CLINICAL TRIAL: NCT03597308
Title: PROSPECTIVE RANDOMIZED CONTROLLED TRIAL COMPARING OXYCODONE, IBUPROFEN AND ACETAMINOPHEN AFTER WIDE AWAKE HAND SURGERY
Brief Title: Prospective Pain Study Comparing Different Treatments After Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018Ilyas
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Opioid Group (Active Comparator)
  Interventions: Drug: 5mg of Oxycodone every 6 hours as needed for pain
- NSAID group (Active Comparator)
  Interventions: Drug: 600mg of Ibuprofen every 6 hours as needed for pain
- Acetaminophen (Active Comparator)
  Interventions: Drug: 500mg of Acetaminophen every 6 hours as needed for pain

INTERVENTIONS:
Drug: 5mg of Oxycodone every 6 hours as needed for pain — 5mg of Oxycodone every 6 hours as needed for pain
  Arms: Opioid Group
Drug: 600mg of Ibuprofen every 6 hours as needed for pain — 600mg of Ibuprofen every 6 hours as needed for pain
  Arms: NSAID group
Drug: 500mg of Acetaminophen every 6 hours as needed for pain — 500mg of Acetaminophen every 6 hours as needed for pain
  Arms: Acetaminophen

SUMMARY:
The purpose of the study is to evaluate the efficacy of three different types of pain medication (Oxycodone - an opioid, Ibuprofen - a non-steroidal anti-inflammatory, and Acetaminophen - a non-opioid analgesic) in the management of postoperative pain following single soft tissue procedures of the hand and wrist performed exclusively under local anesthesia without sedation. The results of this study will help define optimal prescribing guidelines following the two most common hand surgeries while also potentially validating the use of opioid alternatives post-operatively in order to help mitigate excessive or unnecessary dispensal of opioid analgesics.

ELIGIBILITY:
Inclusion Criteria

1. Patients indicated to undergo primary, unilateral carpal tunnel release or trigger finger release surgery under local anesthesia alone.
2. Age eligibility is > 18 years of age.
3. Local anesthesia with 1% lidocaine with 1:100,000 epinephrine and Bicarbonate.

Exclusion Criteria

1. Bilateral procedures.
2. Additional soft tissue or boney procedures performed simultaneously.
3. The use of sedation and/or general anesthesia.
4. Pediatric patients (age < 18 years).
5. Pregnant female patients.
6. Non-English speaking patients.
7. Known allergies or medical contraindications to Oxycodone, Ibuprofen, Acetaminophen.
8. History of chronic pain and/or narcotic use preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Numeric rating Scale for Pain | 2 weeks post-op
  11-point numeric rating scale (NRS) for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No